CLINICAL TRIAL: NCT05289778
Title: Internet Gaming Disorder Among Hong Kong Adolescents: Examining The Socially-Based Intergenerational Transmission Theories
Brief Title: Intergenerational Transmission & IGD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Xue YANG, Research Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 14609820
Record Dates: First submitted 2021-09-29; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Students will complete structured questionnaires in classroom settings, and parents will complete telephone interviews in the absence of their children.

SUMMARY:
This study aims to test the longitudinal association between parental IGD and adolescent IGD, after controlling for covariates at personal, interpersonal and familial levels and the mediation effects of parenting on the intergenerational transmission.

This study is a two-year 3-wave longitudinal study. Students and parents will complete questionnaires at Time1, Time2, and Time3.

DETAILED DESCRIPTION:
Introduction Adolescent Internet Gaming Disorder (IGD) causes severe physical, psychological, and social harms. Family and parents play critical roles in adolescent IGD. Based on the socially-based intergenerational transmission theories, parental IGD may increase the risk of adolescent IGD directly and indirectly.

Objectives The primary objective is to test the longitudinal association between parental IGD and adolescent IGD, after controlling for covariates at personal, interpersonal and familial levels

Subjects and methods This study is a two-year 3-wave longitudinal study. Adolescents will be recruited from Secondary schools using stratified random sampling method. One parent of each adolescent will be invited. Students will finish a set of validated psychological scales in class-room settings, while parents will finish their questionnaires through telephone interviews at Time1, Time2, and Time3.

Outcomes and measures The primary outcome is adolescent IGD symptoms based on DSM-5 IGD symptoms checklist. The secondary outcomes include time spent on Internet-related activities including gaming and gaming attitudes of adolescents.

Data analysis Univariate and multivariate linear/logistic regression analyses will be conducted to test the associations between parental factors (including parental IGD, parental modeling, and parenting practices) and adolescent IGD.

Implications This study will clarify the level of adolescent IGD in Hong Kong to inform policy and planning. It delineates mechanisms concerning intergenerational transmission of adolescent IGD, and shed light on the development of timely and innovative prevention programs based on a family approach and evidence-informed parental training.

ELIGIBILITY:
Inclusion Criteria (adolescent sample):

* Secondary 1-3 students (grade 7-9)
* willingness to finish the study
* Chinese speaking
* living with parent(s)

Inclusion Criteria (parent sample):

* Father or mother of participating child
* living with the participating child
* willingness to finish the study
* Chinese speaking

Exclusion Criteria (adolescent sample):

* receiving treatment for mental disorders
* intellectually disabled

Exclusion Criteria (parent sample):

* lack of competence in the Chinese language
* receiving treatment for mental disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Secondary 1-3 students (grade 7-9) will be recruited from secondary schools using stratified random sampling method. One parent of each student will be invited.
Sampling Method: Probability Sample
Enrollment: 1270 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Adolescent IGD symptoms | 24months
  The DSM-5 classification of IGD: The 9-item IGD checklist is a short, user-friendly, self-report measure for assessing the DSM-5 classification of IGD. Symptoms to be assessed include preoccupation, tolerance, withdrawal, unsuccessful attempts to limit gaming, deception or lies about gaming, loss of interest in other activities, use despite knowledge of harm, use for escape or relief of negative mood, and harm in the past 12 months. Response options are no (0) and yes (1). As per the DSM-5 recommendation, those with >=5 'yes' responses are considered IGD cases. The Chinese version has been validated with high internal consistency.

SECONDARY OUTCOMES:
Time spent on Internet-related activities | 24months
  The China Internet Network Information questionnaire includes 5 items for 5 Internet activities: browsing information and news, playing online games, chatting online, trading online and online entertainment (movies or music) (1=never to 5=always). Number of hours used on different Internet-related activities during a typical week in the last three months will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yang, Principal Investigator — JC School of Public Health and Primary Care, Faculty of Medicine, CUHK
Locations (1):
- Cotton Spinners Association Secondary School, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided